CLINICAL TRIAL: NCT05378555
Title: A Pilot Study of the Use of Oral Ketamine for Treatment of Vaso-Occlusive Pain in Adolescents and Young Adults
Brief Title: Oral Ketamine for Treatment of Vaso-Occlusive Pain
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Christine Greco, Chief, Division of Pain Medicine, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-P00038432
Record Dates: First submitted 2022-04-06; First posted 2022-05-18 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-10

CONDITIONS: Vaso-occlusive Crisis
Keywords: Ketamine; Sickle-cell disease; Opioid-sparing; Analgesia
MeSH Terms: conditions — Vaso-Occlusive Crises; Anemia, Sickle Cell; Agnosia | interventions — Ketamine

STUDY DESIGN:
Intervention Model Description: All patients in this study will receive oral ketamine for the treatment of pain from vaso-occlusive crisis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ketamine (Experimental)
  Interventions: Drug: Ketamine Hydrochloride

INTERVENTIONS:
Drug: Ketamine Hydrochloride — All patients in this study will receive oral ketamine for the treatment of pain from vaso-occlusive crisis. Patients will receive 0.5 mg/kg ketamine Q8hrs for 48 hours.

SUMMARY:
The purpose of this study is to learn more about the feasibility of oral ketamine for the treatment of painful sickle-cell crises in children and adolescents as a supplement to intravenous (IV) opioids. There is a need for improved non-opioid analgesia for patients experiencing sickle-cell crises in the hospital and prehospital setting, as children and adolescents with sickle cell disease who experience sickle-cell crises often have severe pain that is not well controlled by high dose opioids, leading to poor pain management and opioid-related side effects.

The study will begin when patients are admitted to the Emergency Department of Boston Children's Hospital for treatment of a sickle-cell crisis. Oral ketamine will be administered every 8 hours for the next 48 hours. Patients will have continuous cardiorespiratory monitoring for the duration of the study, as per routine care, as well as monitoring by the hospital's Acute Pain Service at least twice daily for pain management and side effects of pain treatment.

At the end of the 48-hour study duration, patients will discuss with the Pain Service and Hematology Service whether to continue oral ketamine, change to intravenous ketamine, or discontinue ketamine based on clinical indications such as level of pain and sedation while on opioids.

DETAILED DESCRIPTION:
This is a pilot study of the feasibility of oral ketamine dosing initiated in the Emergency Department and continued for 48 hours for adolescents and young adults hospitalized with VOCs. A total of 10 patients between the ages of 12 and 24 years will receive oral ketamine 0.5 mg/kg Q8hrs for 48 hours.

Pain scores using VAS and Modified Ramsey Sedation Scores will be obtained every 4 hours per routine nursing care. Vital signs (temperature, heart rate, blood pressure, and respiratory rate) will also be taken every 4 hours throughout the study duration. Side effects (such as dysphoria, dizziness, unpleasant dreams, hallucinations, headache, and nausea) will be monitored throughout the study duration. The Acute Pain Service will assess each patient at least twice daily for pain management and side effects to pain treatment. Ketamine will be discontinued for patients who experience side effects. Patients who experience continued high pain scores will have the option of having oral ketamine discontinued and IV ketamine infusion initiated.

At the end of the 48 hour study period, patient, parent, Pain Service and Hematology Service will discuss whether to continue oral ketamine, change to intravenous ketamine, or discontinue ketamine based on clinical indications such as level of pain and sedation while on opioids. Patients and parents (for patients > 18 years) will be asked to complete a brief satisfaction survey at the end of the 48 hour study period.

Patients who are 12-24 years of age who require admission for vaso-occlusive pain will be included. Patients who do not wish to participate or who have had side effects to previous use of intravenous ketamine for treatment of vaso-occlusive pain that would preclude using ketamine for future pain episodes will not be included in this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients 12-24 years of age who require admission for vaso-occlusive pain

Exclusion Criteria:

* Patients who have had side effects to previous use of intravenous ketamine for treatment of vaso-occlusive pain that would preclude using ketamine for future pain episodes.
* Patient refusal to participate

Ages: 12 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in pain intensity scores using the Visual Analogue Scale (VAS) Pain Score Scale | Baseline, and then every 4 hours for 48 hours
  The Visual Analog Scale (VAS) will be used to measure pain. Scores are recorded on a line that represents a continuum between "no pain" and "worst pain."

SECONDARY OUTCOMES:
Change in Sedation Scores using modified Ramsey Sedation Scores Scale | Baseline, and then every 4 hours for 48 hours
  The Ramsay Sedation Scale used as a measure of sedation allows for a numeric score from 1 to 6, based on responsiveness of the patient. The scale divides a patient's level of sedation into six categories ranging from severe agitation to deep coma.
Number of patients with abnormal vital signs | Baseline, and then every 4 hours for 48 hours
  Vital signs data (blood pressure, heart rate, respiratory rate, and temperature) will be collected and number of patients with abnormal vital signs will be reported.
Frequency of side effects | Baseline, and then every 4 hours for 48 hours
  Side effects such as dysphoria, dizziness, unpleasant dreams, hallucinations, headache, nausea will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ware RE, de Montalembert M, Tshilolo L, Abboud MR. Sickle cell disease. Lancet. 2017 Jul 15;390(10091):311-323. doi: 10.1016/S0140-6736(17)30193-9. Epub 2017 Feb 1. PMID 28159390
- [Background] Neri C, Pestieau S, Young H, Elmi A, et al. Low-dose ketamine for children and adolescents with acute sickle cell disease related pain: a single center experience. J Anesth Clin Res 2014.
- [Background] Telfer P, Kaya B. Optimizing the care model for an uncomplicated acute pain episode in sickle cell disease. Hematology Am Soc Hematol Educ Program. 2017 Dec 8;2017(1):525-533. doi: 10.1182/asheducation-2017.1.525. PMID 29222301
- [Background] Lubega FA, DeSilva MS, Munube D, Nkwine R, Tumukunde J, Agaba PK, Nabukenya MT, Bulamba F, Luggya TS. Low dose ketamine versus morphine for acute severe vaso occlusive pain in children: a randomized controlled trial. Scand J Pain. 2018 Jan 26;18(1):19-27. doi: 10.1515/sjpain-2017-0140. PMID 29794277
- [Background] Hagedorn JM, Monico EC. Ketamine Infusion for Pain Control in Acute Pediatric Sickle Cell Painful Crises. Pediatr Emerg Care. 2019 Jan;35(1):78-79. doi: 10.1097/PEC.0000000000000978. PMID 27902670
- [Background] Bredlau AL, McDermott MP, Adams HR, Dworkin RH, Venuto C, Fisher SG, Dolan JG, Korones DN. Oral ketamine for children with chronic pain: a pilot phase 1 study. J Pediatr. 2013 Jul;163(1):194-200.e1. doi: 10.1016/j.jpeds.2012.12.077. Epub 2013 Feb 10. PMID 23403253
- [Background] Fallon MT, Wilcock A, Kelly CA, Paul J, Lewsley LA, Norrie J, Laird BJA. Oral Ketamine vs Placebo in Patients With Cancer-Related Neuropathic Pain: A Randomized Clinical Trial. JAMA Oncol. 2018 Jun 1;4(6):870-872. doi: 10.1001/jamaoncol.2018.0131. PMID 29621378
- [Background] Rosenblat JD, Carvalho AF, Li M, Lee Y, Subramanieapillai M, McIntyre RS. Oral Ketamine for Depression: A Systematic Review. J Clin Psychiatry. 2019 Apr 16;80(3):18r12475. doi: 10.4088/JCP.18r12475. PMID 30995364